CLINICAL TRIAL: NCT04775823
Title: Evaluation of Hybrid Composite-nanoceramic on Material Characteristic and Clinical Use Over Tooth Wear Patients.
Brief Title: Hybrid Ceramic on Worn Dentition Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201912143RIPB
Record Dates: First submitted 2021-02-16; First posted 2021-03-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Dental Wear
Keywords: Dentistry
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid composite nano-ceramic (Experimental)
  Interventions: Procedure: Hybrid composite nano-ceramic

INTERVENTIONS:
Procedure: Hybrid composite nano-ceramic — Indirect bonding the hybrid composite nano-ceramic restoration to the tooth to be restored of worn dentition patients

SUMMARY:
Evaluation of hybrid composite-nanoceramic on material characteristic and clinical use over tooth wear patients.

DETAILED DESCRIPTION:
Composite resin is often used to restore patient's dental defficiency, and also the material to cover and protect weak tooth structure. In tooth wear patients, multiple factors attributing to destruct their teeth. The durability and strength of the resotrative material must be reinforced. Nanoceramic infiltrated in composite resin may enhance its mechanical characteristics. Therefore, hybrid composite-nanoceramic material may be effective for tooth wear patients.

ELIGIBILITY:
1. Tooth erosion/attrition/abrasion/abfraction patients
2. Age above 20 years old
3. Return at certain period during the trial
4. Full understanding of written and spoken language
5. Agree with the questionnaire

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-02 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the change of hybrid composite-nanoceramic on material characteristic and clinical use over tooth wear patients. | 3months, 6months, 12months, 24months, 36months
  Participants with worn dentition dentition (attrition, erosion, abrasion, abfraction) were enrolled in the present study. They were restored with hybrid composite-nanoceramic resin(Cerasmart, GC Corporation).
  During the follow up time, participants were examined with clinical photos, radiographic film, intraoral scans, and asked to fill in questionnaires. The questionnaires included subjective questionnaire with VAS scale and objective questionnaire according to FDI criteria.
  The restorations were evaluated by two observers at baseline and after 3, 6, 12, 24, 36 months according to the FDI criteria, which were categorized into three groups: esthetic parameters (four criteria), functional parameters (six criteria) and biological parameters (six criteria). Restorations were scored for clinical acceptability. Scores 4 and 5 were recorded as clinically unacceptable, and scores 5 was recorded for clinically failed.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Tsung-Chieh, PhD, Principal Investigator — Associate Professor
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997
- [Result] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Science Committee Project 2/98--FDI World Dental Federation study design (Part I) and criteria for evaluation (Part II) of direct and indirect restorations including onlays and partial crowns. J Adhes Dent. 2007;9 Suppl 1:121-47. PMID 18341239